CLINICAL TRIAL: NCT04023240
Title: 68Ga-FAPI PET Imaging in Malignancy
Brief Title: 68-Ga-FAPI PET Imaging in Malignancy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patients enrolled into study
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-52129; VAR0195 (Other: OnCore)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — 68Ga-FAPI; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI PET/CT (Experimental): Patients receive 68Ga-FAPI IV and then undergo PET/CT approximately 1 hour later.
  Interventions: Drug: 68Ga-FAPI; Procedure: Computed Tomography (CT) scan; Procedure: Positron Emission Tomography (PET) scan

INTERVENTIONS:
Drug: 68Ga-FAPI — 68Ga-FAPI is quinoline based PET radiopharmaceutical.
  68Ga-FAPI is administered intravenously (IV)
  Other Names: 68-Ga-Fibroblast activation protein inhibitor (FAPI)
Procedure: Computed Tomography (CT) scan — Participants will have a CT scan for attenuation correction and anatomic localization of PET data.
Procedure: Positron Emission Tomography (PET) scan — PET images will be acquired.

SUMMARY:
This feasibility trial studies the use of gallium-68 (68Ga)-FAPI as the imaging agent for positron emission tomography (PET)/computed tomography (CT), collectively PET/CT, in patients with various cancers. PET uses a radioactive substance called 68Ga-FAPI, which attaches to cancer activated fibroblasts. The PET scanner takes pictures that capture where the radioactive drug is "lighting up" and attaching to tumor cells, which may help doctors recognize differences between tumor and healthy tissue. CT uses X-rays to make a picture of areas inside the body. Using 68Ga-FAPI in diagnostic procedures, such as PET/CT, may allow doctors to identify smaller tumors than standard imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess feasibility and biodistribution of PET imaging in malignancy using 68Ga-FAPI.

OUTLINE:

Patients receive 68Ga-FAPI intravenously (IV) and then undergo PET/CT approximately 1 hour later.

After completion of study, patients are followed up at 24-72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient with current malignancy confirmed via pathology or imaging
* Patient must be > 18 years old
* Patient must be willing and able to provide written informed consent for the trial
* Patient of reproductive potential will have a pregnancy test

Exclusion Criteria:

* Pregnant or breastfeeding

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-07-14 (Estimated); Study Completion 2023-12-14 (Estimated)

PRIMARY OUTCOMES:
Feasibility of 68Ga-FAPI PET | 24 months
  Feasibility of 68Ga-FAPI PET/CT imaging will be done to assess patients with malignancy. Feasibility will be measured using Likert scale (1-non diagnostic; 5-excellent; anything 3 or more is diagnostic). The study will be feasible if > 50% of scans will have a score of 3 or more

CONTACTS AND LOCATIONS:
Overall Officials: Carina A Mari, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No